CLINICAL TRIAL: NCT05730387
Title: Smart Discharges for Mom & Baby: Saving Mother-newborn Dyads by Developing a Predictive Risk Model to Identify Vulnerable Dyads and Guide Delivery of Evidence-based, Locally-informed Interventions for Targeted Post-discharge Care
Brief Title: Smart Discharges for Mom & Baby
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Matthew Wiens, Assistant Professor, University of British Columbia
Other Study IDs: H21-03709
Record Dates: First submitted 2022-12-09; First posted 2023-02-15 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Maternal Sepsis; Neonatal Sepsis
Keywords: maternal health; neonatal health; patient discharge; post-natal care
MeSH Terms: conditions — Pregnancy Complications, Infectious; Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mother and newborn dyads: We will recruit 6700 mother and newborn dyads from the two participating hospitals. We will continue to follow-up with all patients enrolled in the study until 6 weeks (42 days) post delivery.
  Interventions: Other: Observational only

INTERVENTIONS:
Other: Observational only — This is a non-interventional study

SUMMARY:
This study aims to build a predictive algorithm that identifies mother-newborn dyads most at risk of death or complications in the 6 weeks after birth. The investigators will conduct a multi-site cohort study with 7,000 dyads in Uganda and engage with local stakeholders (e.g., patients, healthcare workers, and health policy-makers) to develop an evidence-based bundle of interventions that address key practice gaps and the critical factors leading to death and complications in these dyads. In the investigator's epidemiological study of post-delivery post-discharge outcomes in 3,236 dyads in Uganda (2017-2020), results indicated that most newborn and maternal readmissions were due to infectious illness (i.e. sepsis, surgical site infections, malaria), and primarily occurred early in the post-discharge period. Thus, the focus of this study will be identifying interventions that target these common and early outcomes, for both mothers and newborns, using World Health Organization recommendations, patient and caregiver experiences, and stakeholder recommendations. If successful, results will inform the next steps of this project, which is the external validation of the model and clinical evaluation of a personalized approach to improving health outcomes and health-seeking behaviour for mothers and newborns.

DETAILED DESCRIPTION:
PURPOSE

Neonatal outcomes are highly correlated with the health of the mother, an example of this is shown repeatedly by poor rates of survival of infants after maternal death. Prediction of risk, based on the mother and infant as a pair, is a major gap in current research and yet vital to the survival of both the mom and the infant. Thus, maternal and child health outcomes can be improved by identifying both mothers and babies at increased risk of mortality or serious morbidity after hospital discharge and allocating scarce resources for targeted follow-up to those most vulnerable. This allows the investigators to not only improve health outcomes but benefits the health system with efficient use of resources.

JUSTIFICATION

Since 2011, the investigators have been working with partners in Uganda to develop, validate, and implement an innovative program for children under 5 years who have been discharged following hospitalization for suspected sepsis. In this research and implementation program, called Smart Discharges, healthcare workers use an individualized risk prediction score to identify children at high risk of death or complications after discharge from a hospital following treatment for suspected sepsis. They can then use this score to guide the intensity of a counselling and community-referral program. While all participants receive counselling, only those above a certain risk threshold receive down-referrals to community health facilities. The investigators have shown that this approach may reduce post-discharge child mortality after in-hospital treatment for suspected sepsis by as much as 30%. Now, the investigators are working to expand their innovative precision public health approach to improving post-discharge care for mother-newborn dyads.

Findings will inform the development an evidence-based bundle of care for both the mother and newborn. This package will ensure that low-risk mother-infant pairs receive less burdensome (yet pragmatic and feasible) postpartum care, while high risk pairs receive a more extensive bundle of interventions (such as education, nutrition, healthcare interaction and community support). The Smart Discharges for Mom & Baby package will include support targeting aspects of both clinical and emotional wellbeing. Additional extensions of this work will include validating the risk models in women who deliver at home or suffer a stillbirth to ensure that more women and babies can benefit from the proposed intervention.

HYPOTHESIS

Maternal and infant characteristics collected at the time of discharge following a facility delivery can predict the risk of maternal or neonatal death or need for re-admission within six weeks of birth.

OBJECTIVE

The primary objective is to inform the development of an integrated maternal and newborn risk-based post-discharge care program. Specifically, the study aims to (1) develop and internally validate clinical risk prediction models for identifying dyads at high-risk of death or hospital readmission in the 6-week post-delivery post-discharge period, and (2) identify gaps and opportunities during in-hospital, discharge, and post-discharge care to inform the future development of an evidence-and risk-based bundle of interventions to improve postnatal care (PNC) for dyads.

DESIGN

This is a mixed-methods study using both quantitative and qualitative techniques to explore and map the current postnatal discharge processes in Uganda using data from two distinct hospital settings.

* Phase I) The team will conduct an observational cohort study informed through direct observation of the mother and newborn dyad prior to facility discharge and after delivery and follow-up telephone interviews conducted at six-weeks post-discharge.
* Phase II) The team will conduct journey mapping with a subset of dyads enrolled in the observational cohort using direct observation and follow-up telephone interviews.
* Phase III) The team will conduct a process mapping exercise using focus group discussion methodology with select facility staff.
* Phase IV) The team will conduct focus group discussions with a subset of mothers enrolled in the observational cohort, as well as their family members.

STATISTICAL ANALYSIS

Quantitative analysis: The investigators will summarize all risk factors for mothers and newborns that do and do not experience poor outcomes and estimate univariate associations. For newborns, data will be reported by sex. Derivation of prediction models will be based on optimization of the area under the receiver operating curve (AUROC) and specificity across a variety of modeling and variable selection approaches (e.g., logistic regression, elastic net, support vector machines). Model performance will be based on appropriate re-sampling techniques for internal validation (e.g., cross-validation, bootstrapping). Focus will be on developing parsimonious predictive models (e.g., 5-10 predictor variables) with high sensitivity (>80%). AUROC, sensitivity, and specificity will be reported for each model, along with positive and negative predictive values. Site specific metrics will be compared to ensure consistency across settings, and re-calibration may be considered if individual site performance is lower than expected. Finally, the investigators will assess combined sensitivity and specificity when each individual model is applied to the dyad. Outside of prediction modelling, the sample size will allow the investigators to detect an odds ratio of at least 1.30 for a given risk factor with 80% power and 5% significance and relative precision of 25%. Statistical analysis of quantitative data from journey mapping observation surveys and patient interviews will be performed using R Statistical software to obtain descriptive statistics of the frequency and distribution of each variable.

Qualitative Analysis: the investigators will analyze data collected descriptively and report summary statistics. A diagram of the discharge process will be developed, identifying key areas for improvement during the peri-discharge and post-discharge process. Focus group discussion data will be analyzed using a framework method, which allows themes to be developed inductively from participants and deductively from existing literature. Through an iterative process, transcripts will be coded and analyzed for descriptive and interpretive themes using NVivo. Descriptive themes include barriers to care and post-discharge health-seeking behaviour, while interpretive themes focus on caregiver perspectives of maternal and neonatal death and the role of the health system. The investigators will generate frequencies to describe reported medical symptoms, health-seeking behaviour, and barriers to care, and summarize common themes. Member checking will be used to improve the validity of the results, creating a summary document of the main findings that will be reviewed by health workers who participated in the focus groups. Feedback from patients and families will be obtained over telephone with research nurses who will explain the main findings verbally.

ELIGIBILITY:
Inclusion Criteria:

* Women and adolescent girls aged 12 and above delivering a single or multiple babies at the study hospital during the active recruitment phase.

Exclusion Criteria:

* Inability, for whatever reason, to provide informed consent.
* Language barrier
* Mother is from a refugee camp
* Mother has no access to phone or other means for follow-up
* Mother lives outside of hospital catchment area

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population represents women living within the catchments of two study hospitals (Mbarara Regional Referral Hospital and Jinja Regional Referral Hospital) in Uganda, who present for delivery.
Sampling Method: Probability Sample
Enrollment: 7182 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew O Wiens, PharmD, PhD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
After the study period, a de-identified copy of the data will be prepared for deposition in a repository with open access with proper governance mechanisms. We will make every effort to prevent re-identification of subjects by coding data that has the potential of being identifiable. For example, we will convert all dates into meaningful decimal numbers (date of birth into days since birth and date of recruitment will be reduced to month of recruitment) and all locations will be coded into data that is useful but not specific (such as address converted to distance and direction from facility). We will ensure that data elements with small numbers of subjects (less than 10) will be coded or lumped to avoid identification. The de-identified study data will be made available using a data hosting service (e.g., Dataverse, Vivli, etc.)
Supporting Information: Study Protocol, SAP
Time Frame: Data will be deposited to an open access repository with moderated access within 2 years of study completion
Access Criteria: Moderated access on a case-by-case basis.

REFERENCES:
- [Derived] Wiens MO, Trawin J, Pillay Y, Nguyen V, Komugisha C, Kenya-Mugisha N, Namala A, Bebell LM, Ansermino JM, Kissoon N, Payne BA, Vidler M, Christoffersen-Deb A, Lavoie PM, Ngonzi J. Prognostic algorithms for post-discharge readmission and mortality among mother-infant dyads: an observational study protocol. Front Epidemiol. 2023 Nov 29;3:1233323. doi: 10.3389/fepid.2023.1233323. eCollection 2023. PMID 38455948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited women presenting for delivery at Jinja and Mbarara Regional Referral Hospitals in Uganda between March 2022 and August 2023 through a quasi-random sampling method. All women enrolled were followed up with, including those who delivered stillbirths or newborns who died in hospital.
Groups:
- Phase I: Observational, Mothers: Mothers were recruited and enrolled from the two participating hospitals and those discharged alive were followed for 6 weeks post-discharge.
- Phase I: Observational, Neonates: Data was collected for all births from the Phase I: Observational, Mothers enrolled in the study, including those that were stillbirths or otherwise dead before being discharged. Follow-up data was only collected for those discharged alive.
Period: Overall Study
Arm/Group | Phase I: Observational, Mothers | Phase I: Observational, Neonates
Started | 7131 | 7359
Discharged | 7129 | 6968
Completed (Participants with a complete six-week follow-up interview) | 7060 | 6891
Not Completed | 71 | 468
Not completed — Stillbirth | 0 | 262
Not completed — Died during or after delivery | 2 | 85
Not completed — Died after being admitted | 0 | 44
Not completed — Lost to Follow-up | 69 | 77

BASELINE CHARACTERISTICS:
Population: Demographics and characteristics of all mothers enrolled (includes two mothers who died giving birth).
Groups:
- Phase I: Observational, Mother: Mother enrolled from the two participating hospitals.
- Phase I: Observational, Neonate: Neonate enrolled after delivery including those that were stillbirths or died before being discharged.
- Total: Total of all reporting groups
Arm/Group | Phase I: Observational, Mother | Phase I: Observational, Neonate | Total
Number analyzed (Participants) | 7131 | 7359 | 14490
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: This measure only applies to mothers. Data for 2 participants (0.03%) is missing.
  years
    number analyzed (Participants) | 7129 | 0 | 7129
    (all) | 26 [22 to 30] |  | 26 [22 to 30]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Neonates: 173 (2.35%) missing
  Participants
    number analyzed (Participants) | 7131 | 7186 | 14317
    Female | 7131 | 3423 | 10554
    Male | 0 | 3763 | 3763
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Lives with the father of the baby [Count of Participants; unit: Participants] — Population: This measure only applies to mothers. Data for 5 participants (0.07%) is missing.
  Participants
    number analyzed (Participants) | 7131 | 0 | 7131
    (all) | 6439 |  | 6439
Education level [Count of Participants; unit: Participants] — Uganda's education system uses a 7-4-2 structure. This consists of 7 years of primary education (P1-P7), 4 years of lower secondary (S1-S4), and 2 years of upper secondary (S5,S6). Population: This measure only applies to mothers. Data for 5 participants (0.07%) is missing.
  Participants
    number analyzed (Participants) | 7126 | 0 | 7126
    ≤ P3 | 263 |  | 263
    P4-P7 | 2263 |  | 2263
    S1-S6 | 3200 |  | 3200
    Post-secondary | 1400 |  | 1400
Transport time [Count of Participants; unit: Participants] — Population: This measure only applies to mothers. Data for 3 participants (0.04%) is missing.
  Participants
    number analyzed (Participants) | 7128 | 0 | 7128
    Less than 30 minutes | 3414 |  | 3414
    30 minutes to 1 hour | 2713 |  | 2713
    >1 hour | 1001 |  | 1001
Had any children who have died [Count of Participants; unit: Participants] — Population: This measure only applies to mothers. Data for 4 participants (0.06%) is missing.
  Participants
    number analyzed (Participants) | 7127 | 0 | 7127
    (all) | 854 |  | 854
Socioeconomic Index Score [Median (Inter-Quartile Range); unit: score on a scale] — This is based on the Global Network Socioeconomic Status Index score that was adapted from the the Multidisciplinary Poverty Index and developed and validated for use in low- and middle-income countries. The scores range from 0 to 10 with a score of 0 to 3 indicating low socioeconomic status (SES), 3 to 6 indicating moderate SES, and 6 to 10 indicating high SES. Population: This measure only applies to mothers. Data for 4 participants (0.06%) is missing.
  score on a scale
    number analyzed (Participants) | 7127 | 0 | 7127
    (all) | 3 [2 to 4] |  | 3 [2 to 4]
Household had sufficient food during pregnancy [Count of Participants; unit: Participants] — Population: This measure only applies to mothers. Data for 5 participants (0.07%) is missing.
  Participants
    number analyzed (Participants) | 7126 | 0 | 7126
    (all) | 1243 |  | 1243
Had admission vitals taken [Count of Participants; unit: Participants] — Population: This measure only applies to mothers. Data for 5 participants (0.07%) is missing.
  Participants
    number analyzed (Participants) | 7126 | 0 | 7126
    (all) | 7020 |  | 7020
Parity [Median (Inter-Quartile Range); unit: pregnancies] — Population: This measure only applies to mothers. Data for 5 participants (0.07%) is missing.
  pregnancies
    number analyzed (Participants) | 7126 | 0 | 7126
    (all) | 2 [1 to 3] |  | 2 [1 to 3]
Diagnosed with chronic illness before pregnancy [Count of Participants; unit: Participants] — Includes HIV, high blood pressure, prior infertility, diabetes, kidney disease, sickle cell, hepatitis B/C, tuberculosis, and chronic mental illness. Population: This measure only applies to mothers. Data for 2 participants (0.03%) is missing.
  Participants
    number analyzed (Participants) | 7129 | 0 | 7129
    (all) | 865 |  | 865
Referral [Count of Participants; unit: Participants] — Population: This measure only applies to mothers. Data for 3 participants (0.04%) is missing.
  Participants
    number analyzed (Participants) | 7128 | 0 | 7128
    (all) | 3163 |  | 3163
Admitted to hospital during pregnancy [Count of Participants; unit: Participants] — Population: This measure only applies to mothers. Data for 4 participants (0.06%) is missing.
  Participants
    number analyzed (Participants) | 7127 | 0 | 7127
    (all) | 1002 |  | 1002
Number of antenatal care visits [Count of Participants; unit: Participants] — Population: This measure only applies to mothers. Data for 4 participants (0.06%) is missing.
  Participants
    number analyzed (Participants) | 7127 | 0 | 7127
    <4 | 1862 |  | 1862
    4-8 | 5140 |  | 5140
    >8 | 125 |  | 125
Diagnosed with a pregnancy-related illness during pregnancy [Count of Participants; unit: Participants] — Includes Gestational diabetes, pre-eclampsia or eclampsia, gestational hypertension, antepartum hemorrhage, PPROM Population: This measure only applies to mothers.
  Participants
    number analyzed (Participants) | 7131 | 0 | 7131
    (all) | 4291 |  | 4291
Mode of Delivery [Count of Participants; unit: Participants] — Population: 3 (0.04%)
  Participants
    number analyzed (Participants) | 7128 | 0 | 7128
    Vaginal | 4546 |  | 4546
    Assisted vaginal | 15 |  | 15
    Caesarean with labour | 1995 |  | 1995
    Caesarean without labour | 572 |  | 572
Surgical urgency of caesarean births [Count of Participants; unit: Participants] — Population: This measure only applies to mothers whose mode of delivery was caesarean. Data for 14 participants (0.55%) is missing.
  Participants
    number analyzed (Participants) | 2553 | 0 | 2553
    Immediate threat to woman or fetus | 1246 |  | 1246
    Maternal/fetal compromise but not immediately life threatening | 877 |  | 877
    Needs early delivery but no maternal/fetal compromise | 30 |  | 30
    At a time to suit the patient and maternity team | 400 |  | 400
Resuscitation at birth [Count of Participants; unit: Participants] — Population: This measure only applies to mothers. Data for 429 participants (6.02%) is missing.
  Participants
    number analyzed (Participants) | 6702 | 0 | 6702
    Not Resuscitated | 4560 |  | 4560
    Resuscitation with oxygen | 265 |  | 265
    Resuscitation without oxygen | 1877 |  | 1877
Number of babies delivered [Count of Participants; unit: Participants] — Population: This measure only applies to mothers. Data for 2 participants (0.03%) is missing.
  Participants
    number analyzed (Participants) | 7129 | 0 | 7129
    Individual | 6907 |  | 6907
    Twin | 217 |  | 217
    Triplet | 5 |  | 5
Mother admitted to higher care following delivery [Count of Participants; unit: Participants] — Population: This measure only applies to mothers. Data for 4 participants (0.06%) is missing.
  Participants
    number analyzed (Participants) | 7127 | 0 | 7127
    (all) | 570 |  | 570
Birth Weight [Median (Inter-Quartile Range); unit: kg] — Population: This measure only applies to neonates. Data for 444 participants (6.03%) is missing. Missing neonate demographics include stillbirths and newborns who died in-hospital.
  kg
    number analyzed (Participants) | 0 | 6915 | 6915
    (all) |  | 3.1 [2.8 to 3.5] | 3.1 [2.8 to 3.5]
Low birthweight (<2500g) [Count of Participants; unit: Participants] — Population: This measure only applies to neonates. Data for 444 participants (6.03%) is missing. Missing neonate demographics include stillbirths and newborns who died in-hospital
  Participants
    number analyzed (Participants) | 0 | 6915 | 6915
    (all) |  | 1038 | 1038
Length [Median (Inter-Quartile Range); unit: cm] — Population: This measure only applies to neonates. Data for 538 participants (7.31%) is missing. Missing neonate demographics include stillbirths and newborns who died in-hospital
  cm
    number analyzed (Participants) | 0 | 6821 | 6821
    (all) |  | 49.5 [48.2 to 50.3] | 49.5 [48.2 to 50.3]
Apgar at 1 minute [Median (Inter-Quartile Range); unit: score] — Apgar score measures the physical health of a newborn shortly after birth. It measures five clinical characteristics: appearance of skin color, heart rate, reflexes, muscle tone, and respiration. Each characteristic is scored from 0 to 2 for a total possible score of 0 to 10, with scores over 7 indicating good health. Population: This measure only applies to neonates. Data for 441 participants (5.99%) is missing. Missing neonate demographics include stillbirths and newborns who died in-hospital
  score
    number analyzed (Participants) | 0 | 6918 | 6918
    (all) |  | 9 [8 to 9] | 9 [8 to 9]
Apgar at 5 minutes [Median (Inter-Quartile Range); unit: score] — Apgar score measures the physical health of a newborn shortly after birth. It measures five clinical characteristics: appearance of skin color, heart rate, reflexes, muscle tone, and respiration. Each characteristic is scored from 0 to 2 for a total possible score of 0 to 10, with scores over 7 indicating good health. Population: This measure only applies to neonates. Data for 441 participants (5.99%) is missing. Missing neonate demographics include stillbirths and newborns who died in-hospital
  score
    number analyzed (Participants) | 0 | 6918 | 6918
    (all) |  | 10 [10 to 10] | 10 [10 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Post-discharge Readmission or Mortality
Description: Composite rate of maternal or neonatal death or re-admission within 6 weeks following delivery
Time Frame: 6 weeks following delivery
Measure: Count of Participants; unit: Participants
Groups:
- Phase I: Observational, Mother: Mother enrolled from the two participating hospitals, survived to discharge and completed the 6-week follow-up
- Phase I: Observational, Neonate: Neonate enrolled after delivery, survived to discharge and completed the 6-week follow-up
Arm/Group | Phase I: Observational, Mother | Phase I: Observational, Neonate
Number analyzed (Participants) | 7060 | 6891
Participants | 231 | 349

2. Secondary Outcome: Post-natal Care Visits
Description: % patients who reported attending at least one post-natal care visits within 6 weeks following delivery
Time Frame: 6 weeks following delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Observational, Mother | Phase I: Observational, Neonate
Number analyzed (Participants) | 7060 | 6968
Participants | 446 | 187

3. Secondary Outcome: Post-discharge Health Seeking
Description: % of patients who reported seeking post-discharge care within 6 weeks following delivery
Time Frame: 6 weeks following delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Observational, Mother | Phase I: Observational, Neonate
Number analyzed (Participants) | 7060 | 6968
Participants
  Care seeking resulted in readmission | 230 | 287
  Care seeking did not result in readmission | 2637 | 1161

ADVERSE EVENTS:
Time Frame: This is an observational study and adverse events are not applicable. All-cause mortality is reported from admission to 6 months post-discharge.
Description: This is an observational study of routine perinatal and neonatal care and no intervention was implemented. Therefore, no Serious or Other Adverse Events were measured/assessed and the population at risk is 0.
  All-cause mortality is reported for all those who were enrolled in the study.
Groups:
- Phase I: Observational, Mother: Mother enrolled from the two participating hospitals and completed the 6-week follow-up
- Phase I: Observational, Neonate: Neonate enrolled after delivery and completed the 6-week follow-up
Arm/Group | Phase I: Observational, Mother | Phase I: Observational, Neonate
All-Cause Mortality (participants affected / at risk) | 3/7131 | 453/7359
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT05730387/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT05730387/ICF_001.pdf